CLINICAL TRIAL: NCT06875960
Title: A Continuation Protocol for Deucravacitinib in Patients With Patients With Systemic Lupus Erythematosus (SLE) or Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE) Who Have Completed Study IM011074 or Study IM011132
Brief Title: A Study to Continue the Administration of Deucravacitinib in Participants With Systemic Lupus Erythematosus (SLE) or Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE) Who Have Completed Study IM011074 or Study IM011132
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-1263
Record Dates: First submitted 2025-03-12; First posted 2025-03-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus (SLE); Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days

SUMMARY:
The purpose of this study is to allow the continued administration of Deucravacitinib in participants with Systemic Lupus Erythematosus (SLE) or Discoid and/or Subacute Cutaneous Lupus Erythematosus (DLE/SCLE) who have completed study IM011074 or Study IM011132

ELIGIBILITY:
Inclusion Criteria

* Participants must have completed Study IM011074 or Study IM011132 through the protocol-required treatment period.
* Participants must be, based on the physician's medical judgement, likely to receive benefit from receiving treatment with deucravacitinib.
* Participants must have received IP within 60 days of enrollment. Exceptions may be granted based upon consultation with BMS.

Exclusion Criteria

* Participants must not have any disease or medical condition that, in the opinion of the physician, would make the subject unsuitable for this protocol, would interfere with the interpretation of subject safety or considered unsuitable by the physician for any other reason.
* Participants must not have any evidence of active Tuberculosis (TB).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated with BMS-986165 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 0001, Farmington, Connecticut
  - New York University School Of Medicine, New York, New York
  - Local Institution - 0003, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06875960.html